CLINICAL TRIAL: NCT00960583
Title: Cost-utility Analysis of a 3-month Exercise Program vs. Routine Follow-up in Patients Having Completed Multidisciplinary Rehabilitation: a Randomized Controlled Trial
Brief Title: Economic Evaluation of an Exercise Program After Multidisciplinary Rehabilitation in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Yves Henchoz, PhD, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIL_PAPA
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Multidisciplinary rehabilitation; Exercise; Cost-effectiveness
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise program (Experimental): Exercise program comprising muscle strengthening, cardiovascular training and stretching exercises.
  Program duration : 12 weeks Sessions frequency : twice per week Session duration : 1h30
  Interventions: Other: Exercise program
- Routine follow-up (Active Comparator): Routine follow-up after functional multidisciplinary rehabilitation by attending physician (Advice to stay active)
  Interventions: Other: Routine follow-up

INTERVENTIONS:
Other: Exercise program — 24 group exercise sessions during 12 weeks
  Arms: Exercise program
Other: Routine follow-up — Advice to stay active
  Arms: Routine follow-up

SUMMARY:
The purpose of the study is to compare, after functional multidisciplinary rehabilitation for chronic low back pain, an exercise program to the routine follow-up which is simply to advice patients to exercise regularly at home. The exercise program should help patients stay active, which should translate into a better long term quality of life and decreased days off work.

ELIGIBILITY:
Inclusion Criteria:

* subacute or chronic low back pain
* phases 2 to 6 of the Krause classification
* without irritative neurological deficit
* age between 18 and 60
* having completed functional multidisciplinary rehabilitation

Exclusion Criteria:

* phases 7 and 8 of the Krause classification
* entitled to a total disability pension
* acute neurological deficit in progress
* sciatica
* pregnancy
* acute inflammatory rheumatic disease
* non-osteoarticular thoracic pain
* spinal fracture within the last 3 months
* osteoporosis
* tumor
* severe heart failure or respiratory failure
* active drug addiction
* current involvement in litigation related to low back pain
* active psychiatric pathology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2005-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | End of functional multidisciplinary rehabilitation, 1 year follow-up
Direct and indirect costs | Before functional multidisciplinary rehabilitation, 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alexander KL So, PhD, FRCP, Study Director — Université de Lausanne, Service de Rhumatologie, Département de l'Appareil Locomoteur, Lausanne, Suisse; Pierre de Goumoëns, MD, Study Chair — Université de Lausanne, Service de Rhumatologie, Département de l'Appareil Locomoteur, Lausanne, Suisse; Michael Norberg, MD, Study Chair — Université de Lausanne, Service de Rhumatologie, Département de l'Appareil Locomoteur, Lausanne, Suisse; Roland Paillex, PT, MS, Study Chair — Centre Hospitalier Universitaire Vaudois (CHUV), Direction des soins, Lausanne, Suisse; Christophe Pinget, PhD, Study Chair — Institute of Health Economics and Management, University of Lausanne and Health Technology Assessment Unit, Medical Direction, University Hospital of Lausanne (CHUV); Jean-Blaise Wasserfallen, MD, MPP, Study Chair — Institute of Health Economics and Management, University of Lausanne and Health Technology Assessment Unit, Medical Direction, University Hospital of Lausanne (CHUV); Yves Henchoz, MS, Principal Investigator — Université de Lausanne, Institut des sciences du sport et de l'éducation physique, Lausanne, Suisse
Locations (1):
- Université de Lausanne, Service de Rhumatologie, Département de l'Appareil Locomoteur, Lausanne, Switzerland

REFERENCES:
- [Result] Henchoz Y, de Goumoens P, Norberg M, Paillex R, So AK. Role of physical exercise in low back pain rehabilitation: a randomized controlled trial of a three-month exercise program in patients who have completed multidisciplinary rehabilitation. Spine (Phila Pa 1976). 2010 May 20;35(12):1192-9. doi: 10.1097/BRS.0b013e3181bf1de9. PMID 20098350
- [Result] Henchoz Y, Pinget C, Wasserfallen JB, Paillex R, de Goumoens P, Norberg M, Kai-Lik So A. Cost-utility analysis of a three-month exercise programme vs usual care following multidisciplinary rehabilitation for chronic low back pain. J Rehabil Med. 2010 Oct;42(9):846-52. doi: 10.2340/16501977-0610. PMID 20878045